CLINICAL TRIAL: NCT02168621
Title: Approaches to Pocket/Root Debridement for Periodontal Infection Control - a Study on Effectiveness.
Brief Title: Intervention Study of Two Protocols for Non-surgical Treatment of Chronic Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGR 2013-2
Record Dates: First submitted 2014-04-10; First posted 2014-06-20 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Non-surgical therapy; Ultrasonic debridement; Scaling and root planing
MeSH Terms: conditions — Chronic Periodontitis | interventions — Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full-mouth ultrasonic debridement (Active Comparator): Motivation and instruction in proper oral hygiene. Before initiation of the subgingival debridement the patient must show sufficient self-performed infection control (full-mouth plaque score <30%). One session of full-mouth ultrasonic pocket/root debridement using a piezoceramic ultrasonic instrument. A follow-up visit after 2-4 weeks is scheduled for oral hygiene control and re-motivation/re-instruction if indicated. At 3 and 6 months re-evaluation is performed and re-instrumentation of all sites showing a remaining probing pocket depth of ≥5 mm carried out. Final evaluation at 18 months.
  Interventions: Procedure: Full-mouth ultrasonic debridement
- Section-wise scaling and root planing (Active Comparator): Conventional treatment approach comprising motivation, oral hygiene instructions and section-wise scaling and root planing at required number of consecutive appointments with 1-2 week interval. Follow-up 2-4 weeks after the last session of SRP for oral hygiene control and re-instruction if indicated. At 3 and 6 months re-evaluation is performed and re-instrumentation of all sites showing a remaining pocket depth of ≥5 mm carried out. Final evaluation at 18 months.
  Interventions: Procedure: Section-wise scaling and root planing

INTERVENTIONS:
Procedure: Full-mouth ultrasonic debridement — Motivation and instruction in proper oral hygiene. Before initiation of the subgingival debridement the patient must show sufficient self-performed infection control (full-mouth plaque score <30%). One session of full-mouth ultrasonic pocket/root debridement using a piezoceramic ultrasonic instrument.
  Arms: Full-mouth ultrasonic debridement
Procedure: Section-wise scaling and root planing — Conventional treatment approach comprising motivation, oral hygiene instructions and section-wise scaling and root planing at required number of consecutive appointments with 1-2 week interval.
  Arms: Section-wise scaling and root planing

SUMMARY:
Treatment directed towards the control of periodontal infections is to about 90% non-surgical procedures. There is evidence from a large number of randomized controlled studies that the efficacy in terms of clinical outcomes of a full-mouth ultrasonic debridement approach (FMUD) is comparable to that of traditional section-wise scaling and root planing (SRP). A hypothesis for the current effectiveness study is that comparable clinical effects will be obtained with the FMUD approach as with conventional section-wise SRP, but with significantly more favourable patient-centred and health-economic outcomes.

This randomized study involves about 100 professionals (dental hygienists) and more than 850 patients at 40 dental clinics in the Vastra Gotaland Region, Sweden. The project not only evaluate treatment effects in terms of pertinent clinical outcomes, it also has a strong focus on patient-centered measures - patient-reported experience measures (PREM) and patient-reported outcome measures (PROM) - as well as health-economics.

DETAILED DESCRIPTION:
All patients with chronic periodontitis (age 30 years and older) attending the selected Public Dental clinics in VG are eligible. The patients should have at least 8 teeth with pathological pockets (probing pocket depth ≥5 mm and bleeding on probing). Only patients providing signed informed consent are included.

Reported data in the study by Wennström et al. (J Clin Periodontol 2005) were used for power calculation. Thus, a total sample of 834 patients will provide a power of 95% at a significance level of p<0.05 to detect a difference of 5% in proportion of sites with "pocket closure" i.e. PPD ≤4 mm and BoP negative (primary efficacy variable) between treatment groups. For a power of 80% a total sample of 506 patients is required.

ELIGIBILITY:
Inclusion Criteria:

* chronic periodontitis
* at least 6 teeth with approximal probing pocket depth ≥5 mm and bleeding on probing

Exclusion Criteria:

* subgingival instrumentation within 6 months prior to screening examination
* compromised medical conditions requiring prophylactic antibiotic coverage

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2014-02; Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
"Periodontal pocket closure" | Up to 18 months
  Frequency of sites with probing pocket depth (PPD) ≤4 mm and no bleeding

SECONDARY OUTCOMES:
Probing pocket depth | Up to 18 months
  Reduction in mean Probing pocket depth
Bleeding on pocket probing (BoP) | Up to 18 months
  Reduction in frequency of bleeding on pocket probing (BoP)
Patient-reported outcome measures (PROM) | Up to 18 months
  Questionnaire
Patient-reported experience measures (PREM) | Up to 18 months
  Questionnaire
Investment for treatment | Up to 18 months
  Individual investment for treatment - Direct and subsidiary costs

OTHER OUTCOMES:
Plaque score | Up to 18 months
  Percentage of tooth surfaces with bacterial deposits
Treatment time | Up to 18 months
  Treatment time in minutes for mechanical instrumentation and oral hygiene instructions respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jan L Wennstrom, Principal Investigator — Dept of periodontology, Sahlgrenska academy, University of Gothenburg, Sweden; Maria Welander, Study Director — Dept of periodontology, Sahlgrenska academy, University of Gothenburg, Sweden; Kajsa H Abrahamsson, Study Director — Dept of periodontology, Sahlgrenska academy, University of Gothenburg, Sweden
Locations (1):
- Dept of periodontology, Institute of odontology, The Sahlgrenska academy at University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Tomasi C, Liss A, Welander M, Alian AY, Abrahamsson KH, Wennstrom JL. A randomized multi-centre study on the effectiveness of non-surgical periodontal therapy in general practice. J Clin Periodontol. 2022 Nov;49(11):1092-1105. doi: 10.1111/jcpe.13703. Epub 2022 Jul 27. PMID 35833528
- [Derived] Liss A, Wennstrom JL, Welander M, Tomasi C, Petzold M, Abrahamsson KH. Patient-reported experiences and outcomes following two different approaches for non-surgical periodontal treatment: a randomized field study. BMC Oral Health. 2021 Dec 15;21(1):645. doi: 10.1186/s12903-021-02001-4. PMID 34911530